CLINICAL TRIAL: NCT02170831
Title: Safety, Pharmacodynamics, and Pharmacokinetics After Multiple Oral Doses of 50, 100, 200, and 400 mg BIBR 1048 MS Solution Administered TID for 7 Days to Healthy Volunteer Subjects. An Open Study, Placebo-controlled Randomised Double Blind at Each Dose Level
Brief Title: Multiple Oral Doses of BIBR 1048 MS Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.2
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (5):
- BIBR 1048 MS low dose (Experimental)
  Interventions: Drug: BIBR 1048 MS low
- BIBR 1048 MS medium dose 1 (Experimental)
  Interventions: Drug: BIBR 1048 MS medium 1
- BIBR 1048 MS medium dose 2 (Experimental)
  Interventions: Drug: BIBR 1048 MS medium 2
- BIBR 1048 MS high dose (Experimental)
  Interventions: Drug: BIBR 1048 MS high
- BIBR 1048 Placebo (Placebo Comparator)
  Interventions: Drug: BIBR 1048 MS placebo

INTERVENTIONS:
Drug: BIBR 1048 MS low
  Arms: BIBR 1048 MS low dose
Drug: BIBR 1048 MS medium 1
  Arms: BIBR 1048 MS medium dose 1
Drug: BIBR 1048 MS medium 2
  Arms: BIBR 1048 MS medium dose 2
Drug: BIBR 1048 MS high
  Arms: BIBR 1048 MS high dose
Drug: BIBR 1048 MS placebo
  Arms: BIBR 1048 Placebo

SUMMARY:
To assess safety, pharmacokinetics and the effect of BIBR 1048 MS on coagulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 45 years
* Broca ≥ -20% and ≤ +20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 1999-05; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Change in aPTT (activated partial thromboplastin time) | up to day 10
Change in PT (prothrombin time) | up to day 10

SECONDARY OUTCOMES:
Cmax (maximum measured concentration) of BIBR 953 ZW | up to day 10
tmax (time from dosing to the maximum concentration) of BIBR 953 ZW | up to day 10
AUC0-∞ (area under the concentration-time curve the time interval from 0 extrapolated to infinity) of BIBR 953 ZW | up to day 10
Cmax,ss (maximum measured concentration at steady state) of BIBR 953 ZW | Day 7
Cmin,ss (minimum measured concentration at steady state) of BIBR 953 ZW | Day 7
Cavg (average plasma concentration at steady state) of BIBR 953 ZW | up to day 10
PTF (percent peak trough fluctuation for the last dosing interval) of BIBR 953 ZW | up to day 10
tmax,ss (time to reach Cmax) of BIBR 953 ZW | up to day 10
t1/2 (terminal half-life) of BIBR 953 ZW | up to day 10
AUCss (area under the plasma concentration-time curve of one dosing interval at steady state) of BIBR 953 ZW | up to day 10
MRTss (mean residence time at steady state) of BIBR 953 ZW | up to day 10
CLtot/F (total apparent clearance) of BIBR 953 ZW | up to day 10
Vz/F (apparent volume of distribution) of BIBR 953 ZW | up to day 10